CLINICAL TRIAL: NCT03223545
Title: Stress Management to Support Women's Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-00725
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Hypertension; Stress; Cardiovascular Diseases
Keywords: mindfulness-based cognitive therapy; Meditation
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based cognitive therapy delivered by telephone (Experimental)
  Interventions: Behavioral: MBCT-T
- Usual Care (UC) (Placebo Comparator)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: MBCT-T — This 8-week program combines mindfulness training with cognitive therapy and is delivered to small groups of patients by telephone using a conference line. Each weekly session is 1 hour long and is comprised of a check-in period, teaching on the week's topic, group discussion, a skill-building exercise, and a home-based practice assignment.
  Arms: Mindfulness-based cognitive therapy delivered by telephone
Behavioral: Usual Care — Treatment guidelines recommend counseling patients with prehypertension on the importance of lifestyle modification to reduce BP. Because of variability in counseling across primary care practices, the study team will provide all participants with NHLBI print educational materials to ensure exposure to lifestyle recommendations: "Your Guide to Lowering Blood Pressure"; and "Facts about the DASH Eating Plan".
  Arms: Usual Care (UC)

SUMMARY:
The purpose of this study is to evaluate a mindfulness-based cognitive therapy intervention delivered over the phone (MBCT-T) for women with prehypertension. MBCT-T is an evidence-based program that teaches meditation practices and cognitive strategies to reduce stress and negative emotions. It targets psychosocial risk factors that disproportionately affect women, including rumination (i.e., negative thinking) and low social support. Investigators plan to translate the established MBCT-T program into Spanish, conduct focus groups to inform cultural adaptations that may be needed for Latina women, and run a pilot randomized controlled trial to test the feasibility, acceptability and effects of MBCT-T on blood pressure and perceived stress in diverse women with prehypertension.

DETAILED DESCRIPTION:
Chronic stress is associated with the development of hypertension and cardiovascular disease. Reducing stress may be a useful prevention strategy for people at elevated risk of hypertension, including those with prehypertension. Women report different types of stress than men and may need tailored stress management programs.

ELIGIBILITY:
Inclusion Criteria:

* Female
* English- or Spanish-speaking
* A current patient of NYU/Bellevue Hospital Center (BHC) for the NYU study site or San Ysidro Health Center (SYHC) for the UCSD study site
* BP measurement in prehypertensive range (SBP 120-139 mmHg or DBP 80-89 mmHg) recorded in EHR within past 6 months AND BP in prehypertensive range at screening
* Willing to provide informed consent and comply with all aspects of the protocol
* Willing to be audio-taped

Exclusion Criteria:

* Current use of antihypertensive medication
* Clinically significant depressive symptoms (PHQ-8 ≥10)
* Significant cognitive impairment, in the EHR or apparent during screening
* History of current diagnosis of schizophrenia or other psychotic disorders
* Current participation in another clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on the study aims, the sample will be 100% female.
Enrollment: 106 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 3 Months
  The mean of three BP readings taken by a trained RA with an automated and validated BP monitor (Microlife WatchBP Office) will be recorded at each visit. Participants will be seated comfortably for 5 minutes with feet flat on the ground prior to measurements. The device will take three readings at 2-minute intervals.

SECONDARY OUTCOMES:
Perceived stress | 3 Months
  Items are rated on a 5-point scale, and higher total scores indicate greater perceived stress.
Measure of Depressive Symptoms using the PHQ-8 | 3 Months
  The PHQ-8 is a validated measure of depressive symptoms during the prior two weeks based on DSM-IV diagnostic criteria for major depression. The PHQ-8 will be completed at screening; patients with scores ≥10, suggestive of clinically significant depressive symptoms, will be excluded and provided with treatment referrals.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Spruill, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States